CLINICAL TRIAL: NCT03117491
Title: Effect of Inferior Alveolar and Gow-Gates Nerve Block Techniques for Symptomatic Mandibular Molars
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Masoud Saatchi, DDS MSc, Professor of Endodontics, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 395437
Record Dates: First submitted 2017-04-03; First posted 2017-04-18 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-04

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: Gow-Gates nerve block; Inferior alveolar nerve block; local anesthesia; molar; pulpitis
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- GGNB injection technique (Active Comparator): In GGNB group, every patient received two1.8-mL cartridges of 2% lidocaine with 1:80,000 epinephrine using the GGNB technique
  Interventions: Procedure: GGNB injections
- IANB injection technique (Active Comparator): In IANB group, every patient received two 1.8-mL cartridges of 2% lidocaine with 1:80,000 epinephrine using the IANB technique
  Interventions: Procedure: IANB injections
- GGNB + IANB injection technique (Active Comparator): In IANB + GGNB group, every patient received one 1.8-mL cartridges of 2% lidocaine with 1:80,000 epinephrine using the IANB technique and one 1.8-mL cartridges of 2% lidocaine with 1:80,000 epinephrine using the GGNB technique
  Interventions: Procedure: GGNB + IANB injections

INTERVENTIONS:
Procedure: GGNB injections — The patients received two GGNB injections of 1.8 mL 2% lidocaine with 1:100,000 epinephrine
  Arms: GGNB injection technique
Procedure: IANB injections — The patients received two IANB injections of 1.8 mL 2% lidocaine with 1:100,000 epinephrine
  Arms: IANB injection technique
Procedure: GGNB + IANB injections — The patients received one GGNB injection plus one IANB injection of 1.8 mL 2% lidocaine with 1:100,000 epinephrine
  Arms: GGNB + IANB injection technique

SUMMARY:
Introduction: to evaluate the efficacy of inferior alveolar nerve block (IANB), Gow-Gates nerve block (GGNB), and their combination in patients with irreversible pulpitis. Methods: One hundred fifty subjects with irreversible pulpitis of a mandibular molar were selected. subjects randomly received two IANB injections or two GGNB injections or their combination of 1.8 mL 2% lidocaine with 1:100,000 epinephrine. Success was specified as no or mild pain on the basis of Heft-Parker visual analogue scale recordings up on the access cavity preparation or initial instrumentation. Data were analyzed by Kruskal-Wallis, and ANOVA tests.

DETAILED DESCRIPTION:
Introduction: to evaluate the efficacy of inferior alveolar nerve block (IANB), Gow-Gates nerve block (GGNB), and their combination in patients with irreversible pulpitis. Methods: One hundred fifty subjects with irreversible pulpitis of a mandibular molar were selected. subjects randomly received two IANB injections or two GGNB injections or their combination of 1.8 mL 2% lidocaine with 1:100,000 epinephrine. Success was specified as no or mild pain on the basis of Heft-Parker visual analogue scale recordings up on the access cavity preparation or initial instrumentation. Data were analyzed by Kruskal-Wallis, and ANOVA tests.

ELIGIBILITY:
Inclusion Criteria:

* vital mandibular molar tooth
* diagnosis of symptomatic irreversible pulpitis

Exclusion Criteria:

* younger than 18 years old
* history of significant medical conditions
* allergies to local anesthetics or sulfites
* pregnancy
* taking any medications that might influence anesthetic assessment
* active sites of pathosis in area of injection
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
the success rate of GGNB local anesthesia technique based on Heft-Parker visual analog scale | at time of access cavity preparation
the success rate of IANB local anesthesia technique based on Heft-Parker visual analog scale | at time of access cavity preparation
the success rate of GGNB + IANB local anesthesia techniques based on Heft-Parker visual analog scale | at time of access cavity preparation

SECONDARY OUTCOMES:
initial pain based on Heft-Parker visual analog scale | before treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No